CLINICAL TRIAL: NCT04171895
Title: Communication Training for Caregivers to Promote Advanced Care Planning
Brief Title: Communication Training for Caregivers In Advanced Care Planning
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-398
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Primary Malignant Brain Tumors; Advanced Care Planning
Keywords: Communication training; 19-398
MeSH Terms: conditions — Brain Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enhanced Usual Care (EUC)
  Interventions: Other: Questionnaires; Other: Enhanced usual care
- Communication Training
  Interventions: Other: Questionnaires; Other: Communication training Part 1 (no longer recruiting); Other: Communication training Part II

INTERVENTIONS:
Other: Questionnaires — Will be filled out before and after the training so investigators can evaluate the skills learned and how they can be used them in advanced care planning. Questionnaires will be available in both paper form and electronic via REDCap.
Other: Communication training Part 1 (no longer recruiting) — 1.5 hour Communication Training will be delivered through videoconferencing using the WebEx or Zoom platforms. The Training consists of a 30-minute lecture watched independently, and two modules (ACP Discussions with your Loved One and ACP Discussions with the Medical Team) completed as part of a virtual meeting. The lecture will be pre-recorded by Drs. Applebaum and Parker and will be sent via REDCap to ICs prior to the training to watch idependently. REDCap will log when ICs watch the lecture so that study staff know the participant has completed this aspect of the training. For the second part of the training ICs will participate in a virtual meeting for approximately 90 minutes of experiential role-play exercises where ICs will practice skills in simulated encounters with actors trained to play patients and HCPs.
  Groups: Communication Training
Other: Enhanced usual care — Participant will complete a survey on distress and receive feedback about distress and given a resource packet with support information and targeted referrals based on needs. The participant will also receive a physical or electronic copy of a book entitled "Cancer Caregiving A to Z" published by the American Cancer Society. At the conclusion of their participation in the study, EUC participants will be given access to the pre-training video and Advanced Care Planning forms sent to Communication Training participants.
  Groups: Enhanced Usual Care (EUC)
Other: Communication training Part II — Part II The communication training developed in Part 1 will have two modules (ACP Discussions with your Loved One and ACP Discussions with the Medical Team) and consist of a 20-30 minute lecture and 90 minutes of experiential role-play exercises where ICs will practice skills in simulated encounters with actors trained to play patients and HCPs. Realistic scenarios were created and tailored according to ICs' reported concerns. After training, ICs will be coached through setting a SMART goal related to conducting ACP conversations, which emphasize Specific, Measurable, Attainable, Relevant and Time-bound steps that motivate and direct behavior change. Two weeks post training, a booster phone call will be made to ICs to check progress toward their SMART goal, address barriers with problem-solving and review skills as indicated.
  Groups: Communication Training

SUMMARY:
The purpose of this research study is to develop and test a new communication training to help caregivers communicate more effectively with their loved ones and healthcare professionals about advanced care planning.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

Informal caregivers:

* Current self-reported informal cancer caregivers (IC) to a patient with a primary malignant brain tumor as per clinician judgment or as per EMR
* English fluency: Self-report by participant identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* age ≥ 18
* has access to a computer or smartphone with a webcam and internet connection

Patients:

* English-speaking as per EMR
* Able to provide informed consent, a determination that will be made in assistance with the patient's medical team.

Part II:

Informal caregivers:

* Current self-reported IC to an MSK patient with a (1) primary malignant brain tumor or (2) leptomeningeal metastasis of a solid tumor, as per clinician judgment or as per EMR.
* English fluency: Self-report by identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* Age >18 as per self report
* Access to a computer or smartphone with a webcam and internet connection as per self report

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For Part 1 and 2 participants will be recruited from the MSK Brain Tumor Center (BTC), a multidisciplinary center comprised of faculty from Neurology, Neurosurgery, Radiation Oncology, Radiology and Psychiatry. The study team may also conduct approaches and recruitment over the phone, in situations where clinic recruitment may not be possible. After screening medical records for eligibility, study staff will email the treating clinician for approach approval, and will only proceed to reach out over phone if the clinician provides explicit permission.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
preliminary efficacy | 1 year
  Feasibility criteria will be met if the target number of participants (n=10) complete a training session within the planned timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm